CLINICAL TRIAL: NCT00329927
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Commercially Available Surface Antigen, Inactivated, (Adjuvanted With MF59C.1) Influenza Vaccine, Formulation 2006-2007, When Administered to Elderly Subjects.
Brief Title: Safety and Immunogenicity of a Commercially Available Influenza Vaccine (Formulation 2006/2007) When Administered to Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70P4S; Eudract number; 2006-000610-20
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Influenza
Keywords: Adjuvanted Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Antigens, Surface

INTERVENTIONS:
Biological: Surface Antigen, Inactivated, (Adjuvanted with MF59C.1), form. 2006-07

SUMMARY:
To evaluate the antibody response to each influenza vaccine antigen when administering a single dose to subjects aged 65 years and over

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older

Exclusion Criteria:

* any serious disease such as cancer, autoimmune disease, advanced arteriosclerotic disease or complicated diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure and bleeding diathesis or conditions associated with prolonged bleeding time
* hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine - - history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* known or suspected (or high risk of developing) impairment/alteration of immune function within the past 7 days
* any acute disease or infections requiring systemic antibiotic or antiviral therapy fever within the past 3 days

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Enrollment: 60
Dates: Start 2006-06

PRIMARY OUTCOMES:
CHMP criteria for evaluation of flu vaccines e.g Seroprotection, GMR's and Seroconversion rate at day 21 following vaccination.

SECONDARY OUTCOMES:
Number and percentage of subjects with at least one local reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one systemic reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one adverse event between Day 0 and the study termination visit (Day 21, window: 20-24).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Chair — Novartis Vaccines & Diagnostics
Locations (2):
- Italy (2):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via Dei Vestini, Chieti
  - Ufficio Igiene e Sanità Pubblica di Lanciano, Via S. Spaventa, 37, Lanciano